CLINICAL TRIAL: NCT04673786
Title: A Randomized, Active-Controlled, Double-Blind, Phase 3 Study to Compare the Efficacy and Safety of CT-P43 to Stelara in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Compare the Efficacy and Safety of CT-P43 to Stelara in Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P43 3.1; 2020-001045-39 (EudraCT Number)
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CT-P43 (Experimental): All patients who were initially randomized to the CT-P43 group on Day 1 (Week 0) will continue their treatment with CT-P43 until Week 40.
  Interventions: Biological: CT-P43
- Stelara (Active Comparator): Patients who were initially randomized to Stelara group on Day 1 (Week 0) will be randomized again in a ratio of 1:1 to either continue Stelara or undergo transition to CT-P43 prior to dosing at Week 16. Thereafter, patients will continue their treatment until Week 40.
  Interventions: Biological: CT-P43; Biological: Stelara

INTERVENTIONS:
Biological: CT-P43 — 45mg or 90mg dose subcutaneous administration
Biological: Stelara — 45mg or 90mg dose subcutaneous administration
  Arms: Stelara

SUMMARY:
This study is a randomized, active-controlled, double-blind, phase 3 study to compare the efficacy and safety of CT-P43 to Stelara in patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
CT-P43, containing the active ingredient ustekinumab, is a human IgG1κ monoclonal antibody that is being developed as a biosimilar medicinal product to the reference product, Stelara. The purpose of this study is to demonstrate similar efficacy and safety of CT-P43 and Stelara in patients with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

- Patient has had diagnosis of plaque-type psoriasis for at least 24 weeks.

Exclusion Criteria:

* Patients diagnosed with forms of psoriasis other than plaque-type.
* Patients previously received ustekinumab or a biosimilar of ustekinumab.
* Patient who has allergies to the active substance or any of the excipients of ustekinumab or study drug, or patients with a hypersensitivity to immunoglobulin products or natural rubber and latex.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre, Tartu, Tartu Country, Estonia, Estonia

REFERENCES:
- [Derived] Papp KA, Lebwohl MG, Thaci D, Jaworski J, Kwiek B, Trefler J, Dudek A, Szepietowski JC, Reznichenko N, Narbutt J, Baran W, Kolinek J, Daniluk S, Bartnicka-Maslowska K, Reich A, Andrashko Y, Kim S, Bae Y, Jeon D, Jung J, Lee H, Pyo T, Ko W. Efficacy and Safety of Candidate Biosimilar CT-P43 Versus Originator Ustekinumab in Moderate to Severe Plaque Psoriasis: 28-Week Results of a Randomised, Active-Controlled, Double-Blind, Phase III Study. BioDrugs. 2024 Jan;38(1):121-131. doi: 10.1007/s40259-023-00630-5. Epub 2023 Nov 22. PMID 37991693

RESULTS

PARTICIPANT FLOW:
Groups:
- CT-P43: Treatment Period I: Patients who were initially randomly assigned to CT-P43 45 mg (who weighed ≤100 kg) or 90 mg (who weighed >100 kg) administered subcutaneously in Treatment Period I (at Weeks 0 and 4) based on patient's baseline body weight.
  Treatment Period II: All patients who received CT-P43 during Treatment Period I and continued to receive CT-P43 in Treatment Period II (at Weeks 16, 28 and 40).
- EU-Stelara: Treatment Period I: Patients who were initially randomly assigned to EU-Stelara 45 mg (who weighed ≤100 kg) or 90 mg (who weighed >100 kg) administered subcutaneously in Treatment Period I (at Weeks 0 and 4) based on patient's baseline body weight.
  Treatment Period II: Patients who were initially randomly assigned to EU-Stelara at Day 1 (Week 0) were to continue to receive EU-Stelara in Treatment Period II (at Weeks 16, 28 and 40).
- Switched to CT-P43: Treatment Period I: Not applicable
  Treatment Period II: Patients who received EU-Stelara during Treatment Period I and re-randomized to receive CT-P43 in Treatment Period II (at Weeks 16, 28 and 40).
Period: Treatment Period I (Weeks 0 to 16)
Arm/Group | CT-P43 | EU-Stelara | Switched to CT-P43
Started | 256 | 253 | 0
Completed | 253 | 249 | 0
Not Completed | 3 | 4 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Period: Treatment Period II (Weeks 16 to 52)
Arm/Group | CT-P43 | EU-Stelara | Switched to CT-P43
Started | 253 | 125 (Patients who had administrated EU-Stelara during Treatment Period I were re-randomized in a ratio of 1:1 to continue EU-Stelara or switch to CT-P43.) | 124 (Patients who had administrated EU-Stelara during Treatment Period I were re-randomized in a ratio of 1:1 to continue EU-Stelara or switch to CT-P43.)
Completed | 239 | 122 | 122
Not Completed | 14 | 3 | 2
Not completed — Withdrawal by Subject | 9 | 3 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- CT-P43: Treatment Period I: Patients who were initially randomly assigned to CT-P43 45 mg (who weighed ≤100 kg) or 90 mg (who weighed >100 kg) administered subcutaneously in Treatment Period I (at Weeks 0 and 4) based on patient's baseline body weight.
- EU-Stelara: Treatment Period I: Patients who were initially randomly assigned to EU-Stelara 45 mg (who weighed ≤100 kg) or 90 mg (who weighed >100 kg) administered subcutaneously in Treatment Period I (at Weeks 0 and 4) based on patient's baseline body weight.
- Total: Total of all reporting groups
Arm/Group | CT-P43 | EU-Stelara | Total
Number analyzed (Participants) | 256 | 253 | 509
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (13.00) | 42.2 (12.64) | 42.4 (12.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 80 | 175
  Male | 161 | 173 | 334
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 25 | 23 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 231 | 230 | 461
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Estonia | 5 | 6 | 11
  South Korea | 25 | 23 | 48
  Poland | 189 | 188 | 377
  Ukraine | 37 | 36 | 73

OUTCOME MEASURES:

1. Primary Outcome: The Mean Percent Improvement From Baseline in PASI Score at Week 12
Description: The percent improvement from baseline in Psoriasis Area and Severity Index (PASI) score at Week 12. PASI score can range from 0 (no psoriasis) to 72 (severe psoriasis).
Time Frame: From baseline to Week 12
Population: Modified ITT Set
Measure: Least Squares Mean (Standard Error); unit: percentage of improvement in PASI score
Arm/Group | CT-P43 | EU-Stelara
Number analyzed (Participants) | 256 | 253
percentage of improvement in PASI score | 77.93 (1.771) | 75.89 (1.739)
Statistical Analysis 1: Comparison: CT-P43 vs EU-Stelara; Test type: Equivalence — Predefined equivalence margin: -10% to 10%; ANCOVA; Multiple imputation (MI) with the Missing at random (MAR) assumption was applied; Treatment difference (%) and 90% CI = 2.05, 90% CI 2-sided [-0.23 to 4.32]

2. Secondary Outcome: The PASI Scores at Week 12
Description: The Psoriasis Area and Severity Index (PASI) score at Week 12. PASI score can range from 0 (no psoriasis) to 72 (severe psoriasis).
Time Frame: Week 12
Population: Modified ITT Set (participants analysed at Week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CT-P43 | EU-Stelara
Number analyzed (Participants) | 256 | 248
score on a scale | 2.98 (3.412) | 3.44 (4.362)

3. Secondary Outcome: The Mean Percent Improvement From Baseline in PASI Score Through Week 52
Description: The percent improvement from baseline in Psoriasis Area and Severity Index (PASI) score through Week 52. PASI score can range from 0 (no psoriasis) to 72 (severe psoriasis).
Time Frame: Through Week 52
Population: Modified ITT Set
Measure: Mean (Standard Deviation); unit: percentage of improvement in PASI score
Groups:
- CT-P43 Maintenance: Treatment Period I: Patients who were initially randomly assigned to CT-P43 45 mg (who weighed ≤100 kg) or 90 mg (who weighed >100 kg) administered subcutaneously in Treatment Period I (at Weeks 0 and 4) based on patient's baseline body weight.
  Treatment Period II: All patients who received CT-P43 during Treatment Period I and continued to receive CT-P43 in Treatment Period II (at Weeks 16, 28 and 40).
- EU-Stelara Maintenance: Treatment Period I: Patients who were initially randomly assigned to EU-Stelara 45 mg (who weighed ≤100 kg) or 90 mg (who weighed >100 kg) administered subcutaneously in Treatment Period I (at Weeks 0 and 4) based on patient's baseline body weight.
  Treatment Period II: Patients who were initially randomly assigned to EU-Stelara at Day 1 (Week 0) were to continue to receive EU-Stelara in Treatment Period II (at Weeks 16, 28 and 40).
Arm/Group | CT-P43 Maintenance | EU-Stelara Maintenance | Switched to CT-P43
Number analyzed (Participants) | 242 | 122 | 123
percentage of improvement in PASI score | 93.79 (11.794) | 93.39 (14.947) | 91.58 (13.264)

4. Secondary Outcome: The Number of Patients Achieving PASI 50, PASI 75, PASI 90, and PASI 100 Responses at Week 12
Description: The number of participants achieving at least 50%/75%/90%/100% improvement from baseline in Psoriasis Area and Severity Index (PASI) at Week 12. PASI score can range from 0 (no psoriasis) to 72 (severe psoriasis).
Time Frame: Week 12
Population: Modified ITT Set
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P43 | EU-Stelara
Number analyzed (Participants) | 256 | 253
Participants
  PASI 50 | 247 | 240
  PASI 75 | 212 | 187
  PASI 90 | 129 | 127
  PASI 100 | 47 | 48

5. Secondary Outcome: The Number of Patients With sPGA Score of Clear (0) or Almost Clear (1) at Week 12
Description: The sPGA is a 5-point score ranging from 0 to 4, based on the physician's assessment of the erythema, average thickness, and scaling of all psoriatic lesions at a given time point. The sum of the 3 scales will be divided by 3 to obtain a final sPGA score.
Time Frame: Week 12
Population: Modified ITT Set
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P43 | EU-Stelara
Number analyzed (Participants) | 256 | 253
Participants | 219 | 201

6. Secondary Outcome: The Change From Baseline in Dermatology Life Quality Index (DLQI) Through Week 52
Description: This DLQI is a 10-item patient-reported outcome questionnaire that, in addition to evaluating overall QoL, can be used to assess 6 different aspects that may affect QoL: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. Total scores range from 0 to 30 (less to more impairment).
Time Frame: Through Week 52
Population: Modified ITT set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CT-P43 Maintenance | EU-Stelara Maintenance | Switched to CT-P43
Number analyzed (Participants) | 242 | 122 | 123
score on a scale | -10.5 (7.24) | -8.5 (7.17) | -9.2 (6.93)

ADVERSE EVENTS:
Time Frame: Through 52 weeks
Description: Treatment Period I: Week 0 to Week 16 pre-dose; Treatment Period II: Week 16 to Week 52 (End-of-study visit)
Groups:
- Treatment Period I: CT-P43: Patients who were initially randomly assigned to CT-P43 45 mg (who weighed ≤100 kg) or 90 mg (who weighed >100 kg) administered subcutaneously in Treatment Period I (at Weeks 0 and 4) based on patient's baseline body weight.
- Treatment Period I: EU-Stelara: Patients who were initially randomly assigned to EU-Stelara 45 mg (who weighed ≤100 kg) or 90 mg (who weighed >100 kg) administered subcutaneously in Treatment Period I (at Weeks 0 and 4) based on patient's baseline body weight.
- Treatment II: CT-P43 Maintenance: All patients who received CT-P43 during Treatment Period I and continued to receive CT-P43 in Treatment Period II (at Weeks 16, 28 and 40).
- Treatment Period II: EU-Stelara Maintenance: Patients who were initially randomly assigned to EU-Stelara at Day 1 (Week 0) were to continue to receive EU-Stelara in Treatment Period II (at Weeks 16, 28 and 40).
- Treatment Period II: Switched to CT-P43: Patients who received EU-Stelara during Treatment Period I and re-randomized to receive CT-P43 in Treatment Period II (at Weeks 16, 28 and 40).
Arm/Group | Treatment Period I: CT-P43 | Treatment Period I: EU-Stelara | Treatment II: CT-P43 Maintenance | Treatment Period II: EU-Stelara Maintenance | Treatment Period II: Switched to CT-P43
All-Cause Mortality (participants affected / at risk) | 0/256 | 0/253 | 1/253 | 0/125 | 0/124
Serious Adverse Events (participants affected / at risk) | 4/256 | 4/253 | 5/253 | 3/125 | 2/124
Other Adverse Events (participants affected / at risk) | 14/256 | 20/253 | 35/253 | 25/125 | 28/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period I: CT-P43 (N=256) | Treatment Period I: EU-Stelara (N=253) | Treatment II: CT-P43 Maintenance (N=253) | Treatment Period II: EU-Stelara Maintenance (N=125) | Treatment Period II: Switched to CT-P43 (N=124)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tubular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period I: CT-P43 (N=256) | Treatment Period I: EU-Stelara (N=253) | Treatment II: CT-P43 Maintenance (N=253) | Treatment Period II: EU-Stelara Maintenance (N=125) | Treatment Period II: Switched to CT-P43 (N=124)
COVID-19 (Infections and infestations) | 11 (11) | 12 (12) | 13 (13) | 11 (11) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 8 (8) | 10 (10) | 4 (4) | 7 (8)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 7 (7) | 4 (4) | 4 (4)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 4 (5)

LIMITATIONS AND CAVEATS:
Due to the conflict in Ukraine, sponsor provided guideline for exceptional allowance regarding visit window and study assessments (only EOS visit was affected) in order to ensure patients' safety and the robustness and integrity of data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT04673786/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT04673786/SAP_001.pdf